CLINICAL TRIAL: NCT01656655
Title: Parenting With and Without PTSD: The Effect of Attachment, Symptoms and Posttraumatic Growth
Brief Title: Effect of Post Traumatic Stress Disorder on Parenting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Rena Cooper, Head Outpatient Psychiatry, Hadassah Medical Organization
Other Study IDs: PTSDpar-2-hmo
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: ptsd, parenting
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PTSD group: Patients with PTSD
- Control Group: non PTSD group

SUMMARY:
PTSD affects a wide variety of symptoms, some of which have been shown to disrupt family relationships. This study will examine some of the effects on parenting, from the perspective of the parent with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* ptsd (PSS>15) children under age 18

Exclusion Criteria:

* non ptsd (pss<15) children under age 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with ptsd
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: rena Cooper, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Choose A State, Israel